CLINICAL TRIAL: NCT04080271
Title: Role of Positron Emission Tomography/Computed Tomography in Detecting Bone Metastases in Cancer Patients.
Brief Title: Role of Positron Emission Tomography/ Computed Tomography (PET/CT) and in Bone Metastases.
Acronym: PET/CT
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aalaa Wael Hussein, resident doctor, Assiut University
Other Study IDs: PET/CT in bone metastases
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Bone Metastases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: 18F-FDG PET/CT — 18F-fludeoxyglucose positron emission tomography/computed tomography

SUMMARY:
The aim of this study is to detect bone metastases by PET/CT examination in cancer patients.

DETAILED DESCRIPTION:
Bone is a fertile soil for dissemination of metastatic tumor cells which can cause either osteolytic ( destructive) or osteoblastic (sclerotic) or mixed lesions in advanced cancer. Bone metastases are most common throughout the axial skeleton, this leads to major complications referred to as skeletal-related events (SREs), the most frequently are the need for radiotherapy and pathological fractures, associated with increase life morbidity and decrease overall survival.

Seeking accurate image modalities provides definite staging, determining the optimal strategy of treatment and precise evaluation to decrease the burden of complication.

PET/CT is superior than 2-dimensional planar providing a better image quality and enables quantitation of tumor metabolism. Acquisition and fusion of PET with CT also allow for localization and morphologic evaluation of abnormalities, leading to increased specificity. The National Comprehensive Cancer Network (NCCN) guideline recommended PET/CT imaging in cancers with high risk skeletal metastases, PET has advantage than CT in diagnosing osteolytic lesions; but combining PET with CT, increase the detection of osteoblastic lesions.

CT is recommended to evaluate structural integrity in revealing cortical integrity and the extent of structural destruction.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with different types of malignant tumor, suspected or diagnosed to have bone metastases and will do PET/CT examination
* patients diagnosed with different types of malignant tumor, with accidently discovered bone metastases during PET/CT examination.
* patients conscious to provide informed consent.

Exclusion Criteria:

* pregnant women.
* patients with blood sugar > 200 mg/dL.
* patients unable to sleep in a fixed position for 20 minutes.
* severely ill patients who aren't capable of complying with study procedures or comatose patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will recruit patients diagnosed with different types of tumors with wide range of age, suspected or diagnosed to have bone metastases, and referred to nuclear medicine unit to perform PET/CT examination, or resulted in to have bone metastases.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
description of bone metastases detected by PET/CT in cancer patients. | one year
  Analysis of number, type and SUVmax of metastatic bony lesions detected by PET/CT in cancer patients.
compare diagnostic performance of PET/CT, planar bone scintigraphy and SPECT/CT in detecting bone metastases | one year
  compare sensitivity, specificity, PPV,NPV and accuracy

SECONDARY OUTCOMES:
risk benefit of PET/CT examination in cancer patients | one year
  To evaluate risk benefit of PET/CT examination in cancer patients suspected to have bone metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A. Mekkawy, Prof. Dr, Study Chair — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Background] Suva LJ, Washam C, Nicholas RW, Griffin RJ. Bone metastasis: mechanisms and therapeutic opportunities. Nat Rev Endocrinol. 2011 Apr;7(4):208-18. doi: 10.1038/nrendo.2010.227. Epub 2011 Jan 4. PMID 21200394
- [Background] Choi J, Raghavan M. Diagnostic imaging and image-guided therapy of skeletal metastases. Cancer Control. 2012 Apr;19(2):102-12. doi: 10.1177/107327481201900204. PMID 22487972
- [Background] Coleman R, Body JJ, Aapro M, Hadji P, Herrstedt J; ESMO Guidelines Working Group. Bone health in cancer patients: ESMO Clinical Practice Guidelines. Ann Oncol. 2014 Sep;25 Suppl 3:iii124-37. doi: 10.1093/annonc/mdu103. Epub 2014 Apr 29. PMID 24782453
- [Background] Crawford ED, Stone NN, Yu EY, Koo PJ, Freedland SJ, Slovin SF, Gomella LG, Berger ER, Keane TE, Sieber P, Shore ND, Petrylak DP; Prostate Cancer Radiographic Assessments for Detection of Advanced Recurrence (RADAR) Group. Challenges and recommendations for early identification of metastatic disease in prostate cancer. Urology. 2014 Mar;83(3):664-9. doi: 10.1016/j.urology.2013.10.026. Epub 2014 Jan 8. PMID 24411213
- [Background] Rosenthal DI. Radiologic diagnosis of bone metastases. Cancer. 1997 Oct 15;80(8 Suppl):1595-607. doi: 10.1002/(sici)1097-0142(19971015)80:8+3.3.co;2-z. PMID 9362427
- [Background] National Comprehensive Cancer Network (NCCN) Breast Cancer NCCN Practice Guidelines in Oncology. Fort Washington, PA:NCCN. 2014. Ver. 2.